CLINICAL TRIAL: NCT01974934
Title: A 12 Week, Open Label, Efficacy and Safety Study of Desvenlafaxine in the Treatment of Vascular Depression
Brief Title: Efficacy and Safety Study of Desvenlafaxine in the Treatment of Vascular Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hotel-Dieu Grace Healthcare (Other Government)
Responsible Party: Principal Investigator, Dr. Corina Velehorschi, MD, FRPC, Hotel-Dieu Grace Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pristiq-2013
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Vascular Depression
MeSH Terms: conditions — Vascular Depression | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desvenlafaxine Succinate (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate

INTERVENTIONS:
Drug: Desvenlafaxine Succinate
  Other Names: Pristiq

SUMMARY:
To examine the efficacy and safety of treatment with desvenlafaxine for vascular depression. Primary efficacy, as it pertains to depressive symptoms, will be assessed by overall change in symptom severity score from baseline to 12-weeks, measured by the Geriatric Depression Scale. The primary efficacy measure of cognition will be the Montreal Cognitive Assessment and analysis of change between baseline and 12-week scores.

To evaluate the effectiveness of desvenlafaxine as a first-line treatment for vascular depression in a sub-group of patients who have experienced a TIA greater than 6 weeks prior to baseline. Mean differences between baseline and 12-week efficacy measures will be examined within the sub-group.

DETAILED DESCRIPTION:
The trial will involve 30 subjects (N=30). The study population is defined on the basis of the broader concept of vascular depression, but not including post stroke depression (PSD). Vascular depression (VaD) is described in patients of age equal or greater than 60 years with clinical symptoms of MDD, evidence of deep white matter hyperintensities (DWMH) on MRI and cognitive deficits not meeting criteria for dementia (based on a score equal or less than 21 on MMSE and 0.5 on CDR).

Upon completion of a screening assessment subjects will begin treatment with desvenlafaxine. For subjects who are currently prescribed an alternate SSRI or SNRI, they will be titrated off their current medication and begin desvenlafaxine, according to the clinical judgment of the investigator based on proven best practices. All subjects will begin on a dose of 50 mg of desvenlafaxine and after 4 weeks of active treatment may be titrated up to 100 mg daily. At the 8-week visit, individuals assessed as partial-responders, in the judgment of the investigator, may be titrated up to 150 mg daily. Personal clinical experience of the principal investigator has shown desvenlafaxine can be safely increased above a dose of 100 mg daily in partially responsive patients. The decision to titrate is based on a risk benefit analysis, as 150 mg is shown to be effective with limited side effects in younger patient populations. The principal investigator is comfortable with a daily dosage of 150mg and will assess for potential side effects. Blood pressure will be monitored at baseline and every 4 weeks as there is evidence that an increase in these values is more likely with dose escalation. It is estimated that 5-15% of the 30 patients may require 150 mg of desvenlafaxine as partial or non-responders to 100 mg daily. Patients prescribed 150mg desvenlafaxine and requiring downward titration will move to 100mg/d for 7 days, then 50mg/d for 7 days, followed by 50mg every other day for 7 days before discontinuation. Patients prescribed 50mg/d or 100mg/d will undergo similar downward titration prior to study drug discontinuation.

A baseline assessment will be conducted on all subjects, followed by assessments at week 4, 8, and a close out assessment at week 12. Additionally, enrolled subjects will undergo an MRI of the head, unless MRI results within the past 6 weeks can be made available, to confirm the presence or absence of DWMH.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
2. Male or female subject between 60 and 80 years of age, at the time of consent.
3. Diagnosis of Major Depressive Disorder according to DSM-IV-TR at screening.
4. Evidence of DWMH on MRI
5. Cognitive deficits not meeting criteria for dementia (MMSE higher or equal 21, Clinical Dementia Rating CDR=0.5, not meeting criteria on DSM IV TR)
6. Subjects are willing and able to comply with scheduled visits, treatment plan, and other study procedures

Exclusion Criteria:

1. Subjects who have a history of repeated non-compliance with treatment.
2. Subjects with any contraindication(s) to desvenlafaxine, in accordance with product monograph
3. Subjects with known or suspected narrow angle glaucoma
4. Subjects currently being treated with anticoagulants
5. Subjects with known hypertension or uncontrolled diabetes
6. Subjects who meet criteria for an active DSM-IV-TR Axis I diagnosis other than Major Depressive Disorder (Cognitive Disorder NOS is permitted but not dementia)
7. Subjects prescribed any Selective Serotonin Reuptake Inhibitors (SSRIs), Serotonin-Norepinephrine Reuptake inhibitors (SNRIs), or typical or atypical antipsychotic medications other than the medications being studied
8. Subjects with a diagnosis of a psychotic disorder or currently experiencing psychotic symptoms
9. Subjects judged by the investigator as being at significant risk of self-injurious/suicidal or violent/homicidal behavior
10. Subjects who have experienced symptoms of a CVA
11. Subjects with TIAs within the past 6 weeks

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | 12-weeks
  To examine the efficacy and safety of treatment with desvenlafaxine for vascular depression. Primary efficacy, as it pertains to depressive symptoms, will be assessed by overall change in symptom severity score from baseline to 12-weeks, measured by the Geriatric Depression Scale. The primary efficacy measure of cognition will be the Montreal Cognitive Assessment and analysis of change between baseline and 12-week scores.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Velehorschi, MD, Principal Investigator — Hotel-Dieu Grace Healthcare
Locations (1):
- Hotel-Dieu Grace Healthcare, Windsor, Ontario, Canada